CLINICAL TRIAL: NCT02070016
Title: Clinical Applicaitons of Non-Invasive Brain Stimulation for the Treatment of Chronic Pain
Brief Title: Transcranial Magnetic Stimulation for Low Back Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sean Mackey, Chief, Division of Pain Medicine, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 27678
Record Dates: First submitted 2014-02-04; First posted 2014-02-24 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- TMS Parameter Condition 1 first (Experimental): Application of Transcranial Magnetic Stimulation
  Interventions: Device: Transcranial Magnetic Stimulation
- TMS Parameter Condition 2 First (Experimental): Application of Transcranial Magnetic Stimulation
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation

SUMMARY:
The purpose of this study is to test whether non-invasive brain stimulation, such as Transcranial Magnetic Stimulation (TMS) may alleviate pain associated with various chronic pain conditions. We will test various methods of TMS to identify a treatment approach that may reduce the symptoms of chronic pain for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Patient with Chronic Low Back Pain
* Meets minimum pain level criteria
* Ability to perform the experimental Task and Procedures

Exclusion Criteria:

* MRI contraindication if an MRI exam is required per protocol
* TMS Contraindication
* History of a psychological or psychiatric disorder that would interfere with study procedures, at the discretion of the researcher.
* Neurologic illness that would interfere with brain integrity
* Current medical condition or medication use that would interfere with study procedures or data integrity, at the discretion of the researcher.
* Currently pregnant or planning to become pregnant.
* On going legal action or disability claim.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in Average Daily Pain | Baseline Compared to each treatmeant series (at 4 weeks, 8 weeks, and 12 weeks)
  Compared to baseline pain report as provided by Visual Analogue Scale (VAS)
Change in Worst Daily Pain | Baseline Compared to each treatment series (at 4 weeks, 8 weeks, and 12 weeks)
  As compared to baseline worst daily pain report provided on visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States